CLINICAL TRIAL: NCT01223326
Title: A Randomized Controlled Trial of N-acetylcysteine to Reduce Ischemia/Reperfusion Injury in Liver Resection Performed Under Ischemic Preconditioning and Intermittent Portal Triad Clamping
Brief Title: N-acetylcysteine to Reduce Ischemia/Reperfusion Injury in Liver Resection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2003/NAC; PIUNA (Other Grant/Funding Number: Plan de Investigación de la Universidad de Navarra)
Record Dates: First submitted 2010-10-15; First posted 2010-10-19 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2012-06

CONDITIONS: Hepatectomy; Reperfusion Injury
Keywords: Acetylcysteine
MeSH Terms: conditions — Reperfusion Injury | interventions — Acetylcysteine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- N-acetylcysteine (Experimental): Intravenous N-acetylcysteine
  Interventions: Drug: Acetylcysteine (NAC)
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Acetylcysteine (NAC) — NAC 150 mg/Kg; and infusion of 50 mg/kg, from 30 minutes before the ischemia up to 60 minutes later to the reperfusion
  Other Names: Flumil
  Arms: N-acetylcysteine
Drug: Saline — Na Cl 0.9% infusion
  Arms: Placebo

SUMMARY:
Study hypothesis: N-acetylcysteine (NAC) can reduce ischemia/reperfusion injury in liver resection performed under ischemic preconditioning and intermittent portal triad clamping.

DETAILED DESCRIPTION:
One of the most important factors in the pathophysiology of liver dysfunction after hepatic surgery is the cellular damage derived from the interruption of blood flood with reperfusion of the organ. N-acetylcysteine (NAC) has proved beneficial in several conditions involving oxidative damage. This study investigates the effects of NAC to reduce ischemia/reperfusion injury in liver resection performed under ischemic preconditioning and intermittent portal triad clamping.

Methods: 46 ASA II-III patients scheduled to undergo liver resection where randomised to receive NAC (initial dose: 150 mg/Kg; and infusion of 50 mg/kg, from 30 minutes before the ischemia up to 60 minutes later to the reperfusion) or placebo in a phase IV clinical trial. Blood, hepatic and urinary markers were obtained at basal status and 1, 3 and 24 h post final reperfusion.

ELIGIBILITY:
Inclusion Criteria:

* Hepatectomy

Exclusion Criteria:

* ASA 4
* Cirrhosis
* Creatinine > 1.2 mg/dL
* Associate surgery (pancreatic or splenectomy)
* Intraoperative bleeding > 2 L.
* Active infection of inflammatory disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2003-01; Primary Completion 2007-10 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Laboratory results | 24 hours
  Coagulation + cytolysis + cholestasis + lactic acid

SECONDARY OUTCOMES:
Inflammation | 24 hours
  Cytokines, adhesion molecules (P-selectin and ICAM-1) and nuclear factor kappaB (NF-kappaB). Circulating neutrophils/platelets. Oxidative stress of neutrophils and apoptosis.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Monedero, M.D., Ph. D., Study Director — Clinica Universidad de Navarra
Locations (1):
- Clinica Universidad de Navarra, Pamplona, Navarre, Spain